CLINICAL TRIAL: NCT02341170
Title: A Phase III Trial of Hippocampal-sparing Prophylactic Cranial Irradiation (HS-PCI) in Locally Advanced (Stage IIIA/IIIB) Adenocarcinoma of the Lung
Brief Title: HS-PCI in Locally Advanced Adenocarcinoma of the Lung
Acronym: HIPPO-S
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Frederik Wenz, Director, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPPO-S
Record Dates: First submitted 2015-01-07; First posted 2015-01-19 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer; Adenocarcinoma; Lymphatic Metastasis
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HS-PCI (Experimental): Hippocampal-sparing prophylactic cranial irradiation (25 Gy in 10 fractions)
  Interventions: Radiation: HS-PCI
- Observation (No Intervention): Observation

INTERVENTIONS:
Radiation: HS-PCI — Hippocampal-sparing prophylactic cranial irradiation with 25 Gy in 10 fractions
  Arms: HS-PCI

SUMMARY:
The primary aim of this study is evaluate the impact of hippocampal-sparing prophylactic cranial irradiation (HS-PCI) on survival status in patients with nodal-positive (locally advanced) adenocarcinoma by comparing overall survival rates of patients undergoing HS-PCI to that of patients without this intervention. In addition, this study aims to investigate whether HS-PCI is detrimental on neurocognitive function and to evaluate its impact on the patient's quality of life.

DETAILED DESCRIPTION:
Patients with locally advanced non-small cell lung cancer (LA-NSCLC) have an increased risk of developing central nervous system (CNS) metastases during the course of their disease. The brain is the most common site of failure after first-line therapies (independent of combined sequential or consolidation chemotherapy). Recent studies employing multimodal therapy have reported overall brain metastasis rates ranging from 22% to 55%, and the rates for brain as first site of relapse range from 16% to 43%.

Prophylactic cranial irradiation (PCI) results in a 2-3 fold lower incidence of brain metastasis. However, randomized studies have failed to demonstrate improved overall survival (OS) after PCI.

One of the major weaknesses of these trials is the unselected mixed pool of stage III patients (stage III A and B, lymph node status N0 to N2, squamous and non-squamous histology etc.). A broad variety of studies have shown that a certain subset of patients with NSCLC (e.g. cancers with adenocarcinoma histology, multilevel nodal involvement) are at highest risk for brain metastases. Furthermore, the risk for brain metastases appears to be specifically higher in younger patients (age <60 years), although this collective commonly undergoes more frequently chemotherapy and/or more aggressive regimens than elderly patients.

Prevention of CNS metastases, even for LA-NSCLC patients with other sites of failure, will improve quality of life and, for patients controlled extracranially, will improve survival. Meta analyses performed on data from several Radiation Treatment Oncology Group (RTOG) studies have shown that longer survival for patients with LA-NSCLC treated with either radiation alone or radiochemotherapy is associated with an increased incidence of CNS metastases. Although the addition of chemotherapy to radiation therapy reduces extracranial distant metastases and improves survival it does not alter brain relapse rates. Even though the addition of modern targeted therapy using small-molecules or antibodies may further improve the outcome, the CNS remains the most common site of failure under targeted therapy, although no evidence for resistance in histological workups of metastases has been found. This emphasizes the urgent need for treatment directed at chemotherapeutically inaccessible (or dormant) micrometastases that are a priori dispersed within the brain. As the median time for relapse in the CNS is approximately 6 months after first-line therapy, the treatment of micrometastases should be meaningfully initiated even during or shortly after first-line therapy.

Irradiation of the brain does not only bear the risk of inducing acute (partially mass-associated) side effects such as nausea, vomiting and fatigue, but also causes long-term neurocognitive deficits. Although neurocognitive disorders after PCI/Whole brain radiotherapy (WBRT) also have a multifactorial etiology based on a patient's individual medical history (preceding chemotherapy, pre-existing vascular damage e.g. from smoking, local reactions/edema), it is currently believed that they are mostly caused by a loss of neural stem cells in the hippocampal areas. Multipotent and self-renewing neural stem cells are found in the subgranular zone of the adult hippocampus and in the subventricular zone of the lateral ventricles. The hippocampus plays an important role in memory consolidation and emotional learning (contextual fear conditioning). The disruption of neurogenesis in the subgranular zone or damage to the hippocampus can lead to impaired short- and long-term memory, learning and contextual fear conditioning. In line with this, irradiating the brain decreases neurogenesis in the hippocampus which leads to impaired hippocampal-dependent learning and memory.

To prevent radiation-induced loss of neuronal stem cells, hippocampus-sparing (HS) radiation techniques have been developed and efficacy has been demonstrated in the recently published phase II RTOG 0933 study. The trial included patients with brain metastases and a Karnofsky Performance Scale (KPS) of 70%. Following HS-WBRT the patients showed a relative neurocognitive function (NCF) decline of 7% four months after HS-WBRT, which is more than four times less than observed in studies with conventional WBRT (30%; p<0.001).

Since the study was a one-arm study without a control, the reported hippocampal failure rate of 4.5% remains controversially discussed. Multiple studies described the hippocampus and limbic circuit to be a generally rare site of brain metastases in many cancers. NSCLC shows a specifically low rate of hippocampal brain metastasis (2.8% of all brain metastases) and risk modelling revealed a only slightly increased absolute risk (+0.2%) after HS-WBRT. Thus, since in the treatment of NSCLC, the efficient prevention of BM and potential CNS micrometastases is currently outweighed by the associated neurotoxicity and a lack of survival benefit, HS-WBRT may provide a possibility to tip the scale toward prophylactic WBRT, at least for a specific subgroup at high risk.

Radiation regimens for PCI that have influenced patterns of CNS failures in NSCLC have included total doses of 20-36 Gy and fraction sizes of 2-3 Gy. A fraction size of 2 Gy and a total dose of 30 Gy was chosen for the RTOG 0214 study of PCI in LA-NSCLC. This regimen has been shown to decrease CNS metastases from 54% to 13% with no difference in NCF decline in PCI versus non-PCI patients at 4 years. In addition, although there is paucity of clinical data from WBRT with doses in the EQD2 (equivalent dose in 2 Gy fractions) range of 10-20 Gy, a dose-response curve providing a 'best fit' model suggests an only minimal benefit from doses above 30 Gy (EQD2).

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed adenocarcinoma of the lung
2. Clinical Stage III with lymph node stage N1-N3
3. Stable disease or any response after definitive or adjuvant radio(chemo)therapy (defined by local standards)
4. No more than 8 weeks after completion of prior radio(chemo)therapy
5. Any acute/subacute ≥ grade 3 toxicities from previous therapy must have resolved to ≤ grade 2 at the time of study entry
6. Age ≥ 18 years and < 75 years
7. ECOG Performance Status ≤ 1
8. Signed study-specific informed consent prior to study entry.

Exclusion Criteria:

1. Stage III with T4 N0
2. Evidence of progressive disease at the time of study entry
3. Brain or leptomeningeal metastases (cMRI not older than 2 weeks)
4. Evidence of extracranial distant metastatic disease
5. Prior cranial irradiation
6. Patients enrolled in other clinical studies that apply or test lung cancer-directed investigational agents/procedures
7. Patients with synchronous or prior malignancy, other than non-melanomatous skin cancer unless disease free greater than 3 years
8. Pregnant women are ineligible as treatment involves unforeseeable risks to the participant and to the embryo or fetus; patients with childbearing potential must practice appropriate contraception.
9. Patients that are unable to undergo repetitive MRI scans
10. Medical conditions that contra-indicate intensive neurocognitive testing (e.g., history of mental retardation, aphasia of any kind, hearing impairment)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
1-year overall survival rate | 1 year

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
Progression-free survival (PFS) | 1 year
Incidence of brain metastasis | 1 year
Incidence of brain metastases within the hippocampal avoidance volume | 1 year
Adverse events | 1 year
Neurocognitive function (NCF), measured by Verbal Learning Memory Test (VLMT) | 1 year
  Verbal Learning Memory Test (VLMT)
  Barthel Activities of Daily Living (ADL) Index
Quality of Life (QoL), measured by Quality of Life Questionnaires / core and brain module (EORTC-QLQ-C30/BN20) | 1 year
  Quality of Life Questionnaires / core and brain module (EORTC-QLQ-C30/BN20)
Activities of Daily Living (ADL), measured by Barthel Index | 1 year
  Barthel Index

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Wenz, MD, Study Chair — Department of Radiation Oncology, University Medical Centre Mannheim; Frank A. Giordano, MD, Principal Investigator — Department of Radiation Oncology, University Medical Centre Mannheim

REFERENCES:
- [Background] Gondi V, Pugh SL, Tome WA, Caine C, Corn B, Kanner A, Rowley H, Kundapur V, DeNittis A, Greenspoon JN, Konski AA, Bauman GS, Shah S, Shi W, Wendland M, Kachnic L, Mehta MP. Preservation of memory with conformal avoidance of the hippocampal neural stem-cell compartment during whole-brain radiotherapy for brain metastases (RTOG 0933): a phase II multi-institutional trial. J Clin Oncol. 2014 Dec 1;32(34):3810-6. doi: 10.1200/JCO.2014.57.2909. Epub 2014 Oct 27. PMID 25349290
- [Background] Ghia A, Tome WA, Thomas S, Cannon G, Khuntia D, Kuo JS, Mehta MP. Distribution of brain metastases in relation to the hippocampus: implications for neurocognitive functional preservation. Int J Radiat Oncol Biol Phys. 2007 Jul 15;68(4):971-7. doi: 10.1016/j.ijrobp.2007.02.016. Epub 2007 Apr 18. PMID 17446005
- [Background] Harth S, Abo-Madyan Y, Zheng L, Siebenlist K, Herskind C, Wenz F, Giordano FA. Estimation of intracranial failure risk following hippocampal-sparing whole brain radiotherapy. Radiother Oncol. 2013 Oct;109(1):152-8. doi: 10.1016/j.radonc.2013.09.009. Epub 2013 Oct 4. PMID 24100152
- [Background] Gore EM, Bae K, Wong SJ, Sun A, Bonner JA, Schild SE, Gaspar LE, Bogart JA, Werner-Wasik M, Choy H. Phase III comparison of prophylactic cranial irradiation versus observation in patients with locally advanced non-small-cell lung cancer: primary analysis of radiation therapy oncology group study RTOG 0214. J Clin Oncol. 2011 Jan 20;29(3):272-8. doi: 10.1200/JCO.2010.29.1609. Epub 2010 Dec 6. PMID 21135270
- [Background] Giordano FA, Welzel G, Abo-Madyan Y, Wenz F. Potential toxicities of prophylactic cranial irradiation. Transl Lung Cancer Res. 2012 Dec;1(4):254-62. doi: 10.3978/j.issn.2218-6751.2012.10.03. PMID 25806190